CLINICAL TRIAL: NCT04593641
Title: A Pilot Phase 1, Randomized, Double-blind, Placebo-controlled, Parallel Group, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Virology of CT-P59 in Patient With Mild Symptoms of SARS-CoV-2 Infection
Brief Title: This is a Phase 1 Study to Evaluate the Safety,Tolerability and Virology of CT P59 in Patients With Mild Symptoms of Symptoms of Coronavirus Disease (COVID-19)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P59 1.2; 2020-003165-19 (EudraCT Number)
Record Dates: First submitted 2020-10-05; First posted 2020-10-20 (Actual); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — regdanvimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 will receive a dose of CT-P59 or matching placebo (Experimental): Drug: CT-P59
  CT-P59 will be administered
  Drug: Placebo
  Placebo-matching CT-P59
  Interventions: Biological: CT-P59
- Cohort 2 will receive a dose of CT-P59 or matching placebo (Experimental): Drug: CT-P59
  CT-P59 will be administered
  Drug: Placebo
  Placebo-matching CT-P59
  Interventions: Biological: CT-P59
- Cohort 3 will receive a dose of CT-P59 or matching placebo (Experimental): Drug: CT-P59
  CT-P59 will be administered
  Drug: Placebo
  Placebo-matching CT-P59
  Interventions: Biological: CT-P59

INTERVENTIONS:
Biological: CT-P59 — administered

SUMMARY:
This is a Phase I study that randomized, double-blind, Placebo-controlled, Parallel Group, Single Ascending Dose Study to evaluate Safety, Tolerability and Virology of CT-P59 in Patient with Mild Symptoms of Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) Infection.

DETAILED DESCRIPTION:
'CT-P59 is a monoclonal antibody targeted against SARS-CoV-2 spike receptor binding protein as a treatment for SARS CoV 2 infection. CT-P59 is currently being developed by the Sponsor as a potential treatment for SARS-CoV-2 infection. In this study, safety, tolerability and virology of CT-P59 will be evaluated in patient with mild symptoms of SARS-CoV-2 Infection.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be randomized in this study:

1. Adult male or female patient, aged between 18 to 60 years (both inclusive).
2. Patient with laboratory confirmed SARS-CoV-2 infection by Reverse Transcription Polymerase Chain Reaction (RT-PCR) at Screening.
3. Patient has mild conditions meeting all of the following criteria:

   1. Oxygen saturation ≥ 94% on room air.
   2. Not requiring supplemental oxygen.
4. Onset of symptom is no more than 7 days prior to the study drug administration.

Exclusion Criteria:

1. Patient with severe condition meeting one of the following:

1. Respiratory distress with respiratory rate ≥ 30 breaths/min.
2. Requires supplemental oxygen.
3. Experience shock.
4. Complicated with other organs failure, and intensive care unit monitoring treatment is needed by investigator's discretion.
5. Any other conditions suspected of being severe symptoms of SARS-CoV-2 infection, in the opinion of the investigator, including but not limited to radiographic findings in lung.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2021-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Incheon Medical Center, Incheon, South Korea

REFERENCES:
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kim JY, Jang YR, Hong JH, Jung JG, Park JH, Streinu-Cercel A, Streinu-Cercel A, Sandulescu O, Lee SJ, Kim SH, Jung NH, Lee SG, Park JE, Kim MK, Jeon DB, Lee YJ, Kim BS, Lee YM, Kim YS. Safety, Virologic Efficacy, and Pharmacokinetics of CT-P59, a Neutralizing Monoclonal Antibody Against SARS-CoV-2 Spike Receptor-Binding Protein: Two Randomized, Placebo-Controlled, Phase I Studies in Healthy Individuals and Patients With Mild SARS-CoV-2 Infection. Clin Ther. 2021 Oct;43(10):1706-1727. doi: 10.1016/j.clinthera.2021.08.009. Epub 2021 Aug 23. PMID 34551869
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- CT-P59 20 mg/kg: Patients were administered CT-P59 (20 mg/kg) by IV infusion with standard of care on Day 1.
- CT-P59 40 mg/kg: Patients were administered CT-P59 (40 mg/kg) by IV infusion with standard of care on Day 1.
- CT-P59 80 mg/kg: Patients were administered CT-P59 (80 mg/kg) by IV infusion with standard of care on Day 1.
- Placebo: Patients were administered Placebo (same volume as the active dose used for CT-P59 in each cohort) by IV infusion with standard of care on Day 1.
Period: Overall Study
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Started | 5 | 5 | 5 | 3
Completed | 4 | 5 | 5 | 3
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 3 | 18
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 59 [49 to 61] | 51 [25 to 52] | 52 [29 to 59] | 50 [49 to 57] | 52 [25 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 0 | 1 | 7
  Male | 2 | 2 | 5 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 5 | 3 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 0 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 5 | 5 | 2 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 5 | 0 | 0 | 1 | 6
  Romania | 0 | 5 | 5 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With TEAEs
Time Frame: Up to Day 14
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 3 | 4 | 3 | 1

2. Primary Outcome: Number of Patients With Treatment-Emergent Serious Adverse Events (TESAEs)
Time Frame: Up to Day 14
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Patients With Treatment-Emergent Adverse Events of Special Interest (TEAESI; Infusion Related Reactions Including Hypersensitivity/Anaphylactic Reaction)
Time Frame: Up to Day 14
Population: Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Patients With Potential Effects on the Incidence of Antibody-Dependent Enhancement (ADE)
Time Frame: Up to Day 14
Population: Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: The Percentage of Patients With Positive/Negative for Quantitative Polymerase Chain Reaction (qPCR)
Time Frame: At Day 28
Population: Intent-to-Treat (ITT) set.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants
  The number of patients with negative for qPCR | 4 | 4 | 2 | 2
  The number of patients with positive for qPCR | 1 | 1 | 2 | 1
  The number of patients who did not obtain any result for qPCR | 0 | 0 | 1 | 0

6. Secondary Outcome: Duration of Viral Shedding in Nasopharyngeal Swab Specimens for qPCR
Time Frame: Up to Day 28
Population: Intent-to-Treat (ITT) set.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
days | 17.49 (6.891) | 12.50 (10.194) | 18.51 (9.344) | 14.19 (11.879)

7. Secondary Outcome: Area Under the Concentration-time Curve of Viral Titers for qPCR
Time Frame: Up to Day 28
Population: Intent-to-Treat (ITT) set.
Measure: Mean (Standard Deviation); unit: (log10cp/mL)*days
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
(log10cp/mL)*days | 55.45 (15.964) | 41.05 (38.738) | 56.26 (28.358) | 60.26 (60.062)

8. Secondary Outcome: Actual Results and Change From Baseline for Viral Shedding in Nasopharyngeal Swab Specimens for qPCR
Time Frame: Up to Day 28
Population: Intent-to-Treat (ITT) set.
Measure: Mean (Standard Deviation); unit: log10cp/mL
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
log10cp/mL
  Actual results for viral shedding in nasopharyngeal swab specimens for qPCR at Day 28 | 0.382 (0.8542) | 0.452 (1.0107) | 1.008 (1.1665) | 0.637 (1.1027)
  Change from baseline for viral shedding in nasopharyngeal swab specimens for qPCR up to Day 28 | -6.326 (0.9801) | -4.258 (1.8477) | -5.723 (1.6683) | -4.367 (1.0060)

9. Secondary Outcome: Number of Patients With Clinical Recovery
Time Frame: Up to Day 28
Population: Intent-to-Treat (ITT) set.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 5 | 5 | 5 | 2

10. Secondary Outcome: Number of Patients Requiring Supplemental Oxygen
Time Frame: Up to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 3 | 0 | 0 | 1

11. Secondary Outcome: Number of Patients With Intensive Care Unit Transfer
Time Frame: Up to Day 28
Population: Intent-to-Treat (ITT) set.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Mechanical Ventilation
Time Frame: Up to Day 28
Population: Intent-to-Treat (ITT) set.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Patients With All-cause Mortality
Time Frame: Up to Day 28
Population: Intent-to-Treat (ITT) set.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Patients With Hospital Admission
Time Frame: Up to Day 28
Population: Intent-to-Treat (ITT) set.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 0 | 0 | 0 | 1

15. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of CT-P59
Description: The PK parameters were calculated by noncompartmental methods based on the actual sampling time points using Phoenix WinNonlin Version 8.3 (Pharsight, St Louis, Missouri, USA).
Time Frame: Up to Day 90
Population: Pharmacokinetic (PK) set.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
hr*ng/mL | 84538893.8 (10202293.97) | 178065255.1 (16390524.47) | 433826801.0 (112102013.80)

16. Secondary Outcome: Time to Cmax (Tmax) of CT-P59
Description: as for outcome 15
Time Frame: Up to Day 90
Population: Pharmacokinetic (PK) set.
Measure: Median (Full Range); unit: hr
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
hr | 2.500 [1.5 to 2.5] | 2.500 [1.55 to 2.58] | 2.500 [1.53 to 2.53]

17. Secondary Outcome: Dose Normalized AUC0-inf (AUC0-inf/Dose) of CT-P59 (Normalized to Total Body Dose)
Description: as for outcome 15
Time Frame: Up to Day 90
Population: Pharmacokinetic (PK) set.
Measure: Mean (Standard Deviation); unit: hr*ng/mL/mg
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
hr*ng/mL/mg | 62595.7 (7539.48) | 58838.6 (10090.23) | 60936.0 (11969.30)

18. Secondary Outcome: Terminal Half-life (t1/2) of CT-P59
Description: as for outcome 15
Time Frame: Up to Day 90
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
hr | 357.1 (41.06) | 380.8 (25.35) | 496.3 (133.26)

19. Secondary Outcome: Percentage of AUC0-inf Obtained by Extrapolation (%AUCext) of CT-P59
Description: as for outcome 15
Time Frame: Up to Day 90
Measure: Mean (Standard Deviation); unit: Percentage of the extrapolated area
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
Percentage of the extrapolated area | 5.917 (10.073) | 1.242 (0.48091) | 3.953 (2.2905)

20. Secondary Outcome: Terminal Elimination Rate Constant (λz) of CT-P59
Description: as for outcome 15
Time Frame: Up to Day 90
Population: Pharmacokinetic (PK) set.
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
1/hr | 0.00196 (0.00024353) | 0.001827 (0.00012290) | 0.001493 (0.00046237)

21. Secondary Outcome: Total Body Clearance (CL) of CT-P59
Description: as for outcome 15
Time Frame: Up to Day 90
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
mL/hr | 16.18 (2.0775) | 17.46 (3.4120) | 16.86 (2.8482)

22. Secondary Outcome: Volume of Distribution During the Elimination Phase (Vz) of CT-P59
Description: as for outcome 15
Time Frame: Up to Day 90
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
mL | 8351.9 (1676.84) | 9514.7 (1357.53) | 11968.2 (3725.56)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date the patients signed the ICF until end-of-treatment visit (up to Day 90).
Description: Treatment Period: Day 1 to Day 90
Arm/Group | CT-P59 20 mg/kg | CT-P59 40 mg/kg | CT-P59 80 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 3/5 | 4/5 | 3/5 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P59 20 mg/kg (N=5) | CT-P59 40 mg/kg (N=5) | CT-P59 80 mg/kg (N=5) | Placebo (N=3)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT04593641/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT04593641/SAP_001.pdf